CLINICAL TRIAL: NCT06815575
Title: A Two-part Phase 1 Open-label Safety and Pharmacokinetic Study of Intravenous RC220 in Combination With Doxorubicin in Adult Patients With Solid Tumours.
Brief Title: A Safety and Pharmacokinetics Study of RC220 Combined With Doxorubicin in Adult Participants With Solid Tumours.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Race Oncology Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAC-010
Record Dates: First submitted 2025-01-20; First posted 2025-02-07 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Solid Tumours; Advanced Solid Tumours
Keywords: Solid Tumours; Advanced Solid Tumours; Phase 1
MeSH Terms: interventions — Doxorubicin

STUDY DESIGN:
Intervention Model Description: The Part 1 dose escalation part of the study will enrol up to 33 patients, guided by the Bayesian Optimal Interval (BOIN) design. Patients will be enrolled in cohorts of 3 for each of the 5 planned dose level cohorts.
  The Part 2 exploratory dose expansion part will enrol a single cohort of approximately 20 patients with solid tumours who have not previously been treated with an anthracycline. Patients will be treated at the MTCD of RC220 and doxorubicin as identified in Part 1. The sample size and patient population cohort will be confirmed following the interim analysis of safety, and PK data after the last patient in Part 1 completes the dose limiting toxicity (DLT) period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part 1: Dose Escalation (Experimental): Participants will receive increasing doses of RC220 on Day 1 of 21-day monotherapy cycle and in combination with the approved fixed dose of Doxorubicin on Day 1 of 21-day combination therapy cycle.
  Combination treatment repeats every 21-day cycle in the absence of disease progression or unacceptable toxicity.
  The aim is to determine safety, tolerability and maximum tolerated combination dosage level to evaluate in Part 2.
  Interventions: Drug: RC220; Drug: Doxorubicin (Adriamycin)
- Part 2: Dose Expansion (Experimental): Participants will receive the tolerated and appropriate combination dosage of RC220 with doxorubicin on day 1 of the 21-day cycle and treatment repeats in the absence of disease progression or unacceptable toxicity.
  The aim is to provide additional safety and tolerability and potential benefits of the combined dosage.
  Interventions: Drug: RC220; Drug: Doxorubicin (Adriamycin)

INTERVENTIONS:
Drug: RC220 — Administered by intravenous infusion over 60 minutes.
Drug: Doxorubicin (Adriamycin) — 60 mg/m2 administered by intravenous infusion over 10 minutes following adminstration of intravenous RC220 on Day 1 of the combination cycles.
  Other Names: Doxorubicin Hydrochloride; Adriamycin®

SUMMARY:
This is a multi-centre, two-part, open-label, phase 1, first in human study of multiple ascending doses of RC220 bisantrene formulation alone and in combination with fixed dose doxorubicin to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD) in adult patients with advanced solid tumours where an anthracycline may be considered as a treatment option / or is indicated.

The study will consist of Part 1 - dose-escalation, to determine the maximum tolerated combination dose of RC220 with doxorubicin to be evaluated in Part 2 - dose-expansion cohort, in patients with solid tumours that are anthracycline treatment naïve and for whom treatment with doxorubicin is indicated. The objective of Part 2 will be to confirm the safety and tolerability and evaluate the preliminary cardioprotective and anti-tumour efficacy of the maximum tolerated combined dose (MTCD) of RC220 with doxorubicin.

DETAILED DESCRIPTION:
This study is an open-label, Phase 1 dose escalation trial with expansion cohort to investigate the safety, tolerability, pharmacokinetics, pharmacodynamics and preliminary cardioprotective and antitumor activity of RC220 in combination with doxorubicin in patients with advanced solid tumours.

The study is divided into two parts: dose escalation (Part 1), and dose expansion (Part 2).

In Part 1(Dose Escalation), patients will be enrolled sequentially into escalating dose cohorts up to 5 planned dose cohorts. Each patient in a dose cohort will receive an intravenous (IV) infusion of RC220 on Day 1 of the lead-in 21-day cycle and continue to the combination cycle, where patients will receive IV RC220 followed by IV doxorubicin on Day 1 of a 21-day cycle . New patients will be enrolled in each dose escalation cohort based on safety observed during the first 21 days of RC220 and doxorubicin combination treatment Cycle 1 until the MTCD is defined based on the recommendations of the Safety Review Committee (SRC). Patients will continue to be treated beyond the first combination cycle observation period until disease progression, unacceptable toxicity, withdrawal of consent or defined end of study, whichever occurs first.

An interim analysis of the accumulated safety, PK, early efficacy and PD (as available) will be conducted to confirm the MTCD of RC220 in combination with fixed dose doxorubicin for further evaluation of the safety and tolerability, preliminary cardioprotective and anti-tumour efficacy in an exploratory dose expansion cohort of patients with solid tumours that are anthracycline treatment naïve and for whom treatment with doxorubicin is indicated.

ELIGIBILITY:
Inclusion Criteria (For Part 1 and Part 2):

1. Able to give voluntary informed consent and understand the study and are willing to follow and complete all the study required procedures.
2. Aged ≥ 18 years at the time of informed consent.
3. Life expectancy ≥ 3 months.
4. Have measurable or evaluable disease per RECIST v1.1. The target lesions must not have prior radiation or other locally treated area unless imaging-based progression has been clearly documented following radiation or other local therapy.
5. Adequate haematological, liver, and kidney function as follows:

   1. Bone marrow reserve:

      • Absolute neutrophil count (ANC) ≥ 1.5 × 109/L without growth factor support in the 2 weeks prior to study entry.

      • Haemoglobin ≥ 90 g/L without transfusion and/or without growth factor support in 2 weeks prior to study entry.
      * Platelet count ≥ 100 × 109/L without transfusion in 2 weeks prior to study entry.
   2. Hepatic function:

      * Aspartate aminotransferase (AST), alanine aminotransferase (ALT) < 3 × upper limit of normal (ULN) (≤5 × ULN if liver metastases or hepatic cell carcinoma (HCC)).
   3. Renal function:

      * Serum creatinine < 1.5 × ULN or Serum creatinine clearance (CrCL) > 50 mL/min, as per the Cockcroft-Gault Equation Glomerular Filtration Rate: [(140-age in years) × weight in kg] / (7.2 × serum creatinine in mg/dL) (× 0.85 for females).

   In PART 2 only: Out of range values for 5a, b and c are allowable based on the discretion of the Investigator and with approval from Sponsor Medical Monitor.
6. International normalized ratio (INR) /prothrombin time (PT) < 2 x ULN, activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN.

   In PART 2 only: Out of range values are allowable based on the discretion of the Investigator and with approval from Sponsor Medical Monitor.
7. Practice adequate contraceptive measures as per below:

   Female patients must:
   * Be of nonchildbearing potential i.e., surgically sterilised or postmenopausal, or;
   * If of childbearing potential, must have a negative serum pregnancy test at Screening and a negative urine pregnancy test before the first study drug administration and on Day 1 of each Cycle. They must agree not to attempt to become pregnant, must not donate ova, and must agree to use 2 forms of highly effective contraceptive method between signing consent, during the study, and at least 90 days after the last dose of study drug, OR use 1 form of highly effective contraceptive method, plus an additional barrier method of contraception between signing consent, during the study, and at least 90 days after the last dose of study drug.
   * Women of childbearing potential with same sex partners (abstinence from penile vaginal intercourse) are eligible when this is their preferred and usual lifestyle.

   Male patients must:
   * be willing not to donate sperm and if engaging in sexual intercourse with a female partner who could become pregnant, a willingness to use a condom in addition to having the female partner use a highly effective contraceptive method between signing consent, during the study, and at least 90 days after the last dose of the study drug.

   PART 1 only - Dose Escalation Specific Inclusion Criteria
8. Histologically/cytologically confirmed, locally advanced unresectable or metastatic solid tumours for whom prior treatments have failed, and where an anthracycline may be considered as a treatment option or is indicated. Note that certain malignancies can be included based on imaging (e.g., HCC) based on the discretion of the Investigator with Sponsor Medical Monitor approval.
9. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1
10. Adequate Hepatic function as per below:

    * Serum Total bilirubin (TBIL) as per below:

      1. Patients with documented Gilbert's syndrome - baseline TBIL < 3 × ULN,
      2. Patient with either HCC or liver metastases - baseline TBIL < 2 × ULN
      3. All other patients baseline TBIL < 2 × ULN. Exceptions are allowable based on the discretion of the Investigator and with approval from Sponsor Medical Monitor

PART 2 only - Exploratory Dose Expansion Specific Inclusion Criteria 8. Histologically/cytologically confirmed solid tumours of any stage for which the patient has not received prior treatment with an anthracycline and for whom treatment with doxorubicin is indicated.

9. ECOG performance status ≤ 2 10. Adequate Hepatic function as per below:

• Serum TBIL as per below:

1. Patients with documented Gilbert's syndrome - baseline TBIL < 3 × ULN,
2. Patient with either HCC or liver metastases - baseline TBIL < 3 × ULN
3. All other patients baseline TBIL < 2 × ULN. Exceptions are allowable based on the discretion of the Investigator and with approval from Sponsor Medical Monitor

Exclusion Criteria (for Part 1 and Part 2):

1. Females who are pregnant or nursing.
2. Received cancer-directed therapy within the following timeframes:

   1. Antitumour therapy (chemotherapy, antibody therapy, molecular targeted therapy, hormonal therapy or investigational agent) within 28 days prior to the first dose of study treatment (or 5 times the half-life if shorter than 28 days, there can be exceptions on a case-by-case as approved by Sponsor Medical Monitor based on pharmacology). Note: concurrent use of hormone deprivation therapy for hormone-refractory prostate cancer, bisphosphonate or denosumab for skeletal related events per institution guideline is permitted.
   2. Wide-field radiation therapy within 28 days (or palliative radiation therapy within 7 days) prior to the first dose of study treatment or has not recovered from the side effects of radiation therapy in the opinion of the Investigator.
   3. Any other concurrent investigational device(s) or conventional agent(s) within 28 days (unless 5 times the half-life is shorter than 28 days) prior to the first dose of study treatment.
   4. Therapeutic radiopharmaceuticals must be stopped 8 weeks prior to the first dose of the study drug.
3. Persisting Grade 2 or higher severity AEs from prior antitumour treatment as per CTCAE v5.0. Patients with pre-existing non-treatable Grade 2 toxicities may be eligible per discretion of the Investigator and with approval from Sponsor Medical Monitor (e.g., Grade 2 chemotherapy induced neuropathy).
4. Patients with primary central nervous system (CNS) malignancy, symptomatic CNS metastases, meningeal metastases or leptomeningeal disease are not allowed.

   Note: Patients with asymptomatic CNS metastases are eligible if clinically controlled, which is defined as 1) ≥ 4 weeks of stable neurologic function following CNS-directed therapy prior to the first dose of study treatment 2) no evidence of CNS disease progression as determined by radiographic imaging ≥ 4 weeks prior to the first dose of study treatment, 3) ≥ 2 weeks from discontinuation of anti-seizure and steroid therapies (receiving prednisone ≤ 10 mg or equivalent steroid therapies is allowed) prior to the first dose of study treatment.
5. Had major surgery within 28-days of the Screening Visit. Note: Patients who have undergone a non-major surgical procedure within 28-days prior to Screening must have recovered adequately from the surgery before the administration of the first dose of study drug. Exception: no waiting period applies following central venous catheter placement.
6. History of tissue or organ transplantation.
7. Treatment with systemic immunosuppressive medications within 4 weeks prior to the first dose of study drug. Exceptions: Daily prednisone equivalent ≤10 mg/day; topical, inhaled, or intranasal corticosteroids.
8. History of severe infection deemed clinically significant by the Investigator or designee within 4 weeks or signs and symptoms of any active infection within 2 weeks prior to the first dose of study treatment.
9. Active hepatitis B or C. Note: Hepatitis B virus (HBV) carriers without active disease (HBV DNA titer < 1000 copies/mL or 200 IU/mL) or cured hepatitis C (negative HCV RNA test) with confirmed viral clearance that are not receiving ongoing treatment and without residual chronic liver disease may be enrolled.
10. Confirmed human immunodeficiency virus (HIV) infection and receiving anti-retroviral therapy (ART). Patients with well controlled HIV infection (i.e., CD4+ count >350 cells/μL and viral copies less than 400/mL after at least 4 weeks of ART) may be eligible per discretion of the Investigator and with approval from Sponsor Medical Monitor.
11. Patients with any inherited predisposition to bleeding or to thrombosis (von Willebrand disease, haemophilia, etc.). Patients with a history of nontraumatic haemorrhage (i.e., end stage liver disease, any haemorrhage requiring medical intervention), thromboembolic event or any condition which may increase bleeding risk including clotting disorders, thrombocytopenia during the last 3 months prior to the first dose of study drug administration.
12. Receiving immunosuppressive or myelosuppressive medications that would, in the opinion of the Investigator, increase the risk of serious neutropenic complications.
13. Any other disease or clinically significant abnormality in laboratory parameters, including serious medical or psychiatric illness/condition, which in the judgement of the Investigator might compromise the safety of the patient or integrity of the study, interfere with the patient's participation in the trial or compromise the trial objectives.
14. Known allergies, hypersensitivity, or intolerance to the study drug or its excipients.
15. Any known, documented, or suspected history of illicit substance abuse that would preclude patient from participation, unless clinically justified (i.e., will not interfere with study participation and/or will not compromise trial objectives) per judgement of the Investigator and with approval of Study Medical Monitor. Exception: Physician-prescribed medicinal opioids or cannabinoids are allowed for pain management.
16. Vaccinated with any live vaccine within 4 weeks prior to the first dose of study treatment.
17. Judgement by the Investigator that the patient is unlikely to comply with study procedures, restrictions and requirements.
18. Use of prescription or non-prescription medications, including complementary medicines, within 14 days or 5 half-lives (whichever is longer) if the medication is a potential inhibitor of cytochrome P450 (CYP) isoform 3A4 or 2D6, and/or P-glycoprotein (P-gp), or if the medication is an inducer of CYP3A4 or P-gp, prior to dosing and throughout study participation.

    PART 1 only - Dose Escalation Specific Criteria
19. Severe or uncontrolled cardiac disease requiring treatment, CHF (New York Heart Association) NYHA III or IV, unstable angina pectoris even if medically controlled, history of myocardial infarction during the 6 months prior to screening, serious arrhythmias requiring medication (with exception of atrial fibrillation or paroxysmal supraventricular tachycardia).
20. Treatment with prior anthracyclines exceeding the maximum equivalent cumulative lifetime dose. In certain cases, patients who have received total cumulative doses may be considered suitable at the discretion of the Investigator in consultation with the patient and the Sponsor Medical Monitor.

PART 2 only -Dose Expansion Specific Criteria 19. Uncontrolled or severe cardiac disease that in the opinion of the Investigator would prevent treatment with doxorubicin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2025-04-02 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Part 1. Incidence of dose limiting toxicities (DLTs) | During the first cycle of RC220 and doxorubicin treatment (1-21 days)
  Evaluated at each dose level RC220 combined with doxorubicin, as graded by National Cancer Institute (NCI) Common Terminology for Adverse Events (CTCAE) version 5.0.
Part 1 and Part 2. Treatment emergent adverse events (TEAE) and serious adverse events (SAEs), | First dose up to 30 days post last combination dose (up to 12 months)
  This includes clinically significant changes in vital signs, physical examination, electrocardiogram, echocardiogram and clinical laboratory tests, as graded by NCI CTCAE v5.0.

SECONDARY OUTCOMES:
Part 1. Maximum tolerated combined dose (MTCD) | After the first dose of RC220 and doxorubicin treatment cycle (1-21 days)
  The MTCD is based on the incidence of Dose Limiting Toxicities (DLTs).
Part 1. Best Overall Response (BOR) | Up to 12 months
  Percentage of patients with best confirmed overall response of clinical response (CR) or partial response (PR) (evaluated by the investigator according to RECISTv1.1) until the time of disease progression.
Part 1. Duration of Response (DOR) | Up to 12 months
  Defined as the time from the earliest date documented (CR or PR) (evaluated by the investigator according to RECISTv1.1) until disease progression or death (by any cause, in the absence of progression).
Part 1. Progression Free Survival (PFS) | Up to 12 months
  Defined as the time of first treatment until disease progression or death (by any cause, in the absence of progression).
Part 2. Change from baseline in cardiac blood biomarker levels (hs-troponins and NT-proBNP), as measured by laboratory tests | up to 12 months
Part 2. Change from baseline in 2D-echocardiogram measurements including GLS, LV volume, LV mass, transmitral flow, atrial volumes. | Up to 12 months
  2D-echocardiograms are performed at specified timepoints. Each time a 2D-echocardiogram is performed, multiple measures will be collected, aggregated and reported on once by a single observer.
  Measures collected from each 2D-echocardiogram, and compared to baseline, include:
  * global longitudinal strain
  * left ventricular mass
  * left ventricular volumes
  * transmitral flow
  * left atrial volume
Part 2. Change from baseline in cardiac magnetic resonance imaging (cMRI) cardiac function parameters (blood flow, global ventricular function, myocardial perfusion) | Up to 12 months
  Each time a cMRI is performed, cMRI images are collected, assessed, compared and reported on in an aggregated manner by an independent cardiologist for changes in cardiac function measures (blood flow, global ventricular function, myocardial perfusion).
Part 2. Change from baseline in functional volume of peak oxygen uptake (VO2 peak). Defined as the highest amount of oxygen consumed at peak exercise. | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Marinella Messina, Study Director — Race Oncology Ltd
Locations (5):
- Australia (3):
  - Gosford Hospital, Gosford, New South Wales
  - Cancer Care Foundation, Miranda, New South Wales
  - Wyong Hospital, Wyong, New South Wales
- Hong Kong (2):
  - Queen Mary Hospital, Hong Kong
  - Prince of Wales Hospital, Shatin

IPD SHARING:
Plan to Share IPD: Undecided